CLINICAL TRIAL: NCT01532479
Title: Saliva, Hyperbaric Oxygen Therapy, & Gland Function: A Prospective Study
Acronym: SHOTGUN
Status: Withdrawn | Type: Observational
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Other Study IDs: SHTGN-001
Record Dates: First submitted 2012-02-08; First posted 2012-02-14 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Osteoradionecrosis of the Jaw; Xerostomia
Keywords: Osteoradionecrosis; Xerostomia
MeSH Terms: conditions — Xerostomia; Osteoradionecrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Treatment Group: Subjects with ORN treated with Hyperbaric Oxygen Therapy
- Postive Control Group: Subjects treated with Hyperbaric Oxygen Therapy that have not had head or neck radiation therapy
- Negative Control Group: Subjects who have had head and neck radiation that have not had Hyperbaric Oxygen Therapy

SUMMARY:
The purpose of this study is to determine if Hyperbaric Oxygen (HBO) therapy improves salivary gland function in previously head-and-neck irradiated patients. The following will be evaluated: salivary a-amylase, IGF-1, Thrombospondin-1, and VEGF-A concentrations, resting and stimulated salivary flow rate and pH, and salivary buffering capacity. Demographic data, past medical/surgical histories, social history and habits, risk factors, medication list, nutritional status, stage and location of tumor treated, dose/duration of radiation, and time elapsed since radiation treatment will be reviewed and recorded. Subjects will complete a quality of life questionnaire, describe (presence/absence) dry mouth symptoms prior to HBO therapy, and provide current A1c level, or submit to a finger stick. The following groups will be evaluated: 1. Head-and-neck irradiated subjects with ORN (indicating HBO therapy) 2. Subjects with other conditions indicating HBO therapy (positive control), and 3. Head-and-neck irradiated subjects without ORN (negative control). Subjects will include 78 males or females, 18 years old and over. In total, participation will last 22 weeks.

DETAILED DESCRIPTION:
This is a prospective study in a human model examining treatment of patients who have sustained damage to salivary glands following head and neck radiation, subsequent xerostomia, and who are currently indicated for hyperbaric oxygen therapy for treatment of osteoradionecrosis. Salivary flow rates, pH and buffering capacity before and after hyperbaric oxygen treatments will be collected using GC America (Alsip, Illinois) Saliva-Check BUFFER Kit and results will be recorded. The 6 tests take 10 minutes to complete per patient. According to GC America, these tests are simple, demonstrate salivary dysfunction, help identify factors affecting salivary dysfunction, and assist in the diagnosis of xerostomia. Salivary testing and data collection will occur on 8 independent visits over the course of hyperbaric oxygen treatment and during follow-up. Stimulated saliva samples will be used to measure proteins that are involved in salivary gland revascularization and repair. Saliva samples will be stored at less than or equal to -20C for up to 1 year. Measurements of salivary VEGF-A, IGF-1, and Thrombospondin-1 will be quantified using R&D Systems (Minneapolis, MN) ELISA kits and results will be recorded. Salivary Alpha-Amylase will be measured using Rocky Mountain Diagnostics, Inc (Colorado Springs, CO) Alpha-Amylase Saliva kit. Protein analysis will be done on stimulated saliva samples collected at 4 independent visits: first week, fourth week, eighth week, sixteenth week.

The medical, surgical, and health histories of each participant will be reviewed. Each participant will complete the EORTC quality of life core questionnaire (QLQ - C30 v3.0), including head and neck cancer module, at the start and completion of the trial. A blood sample from each participant will be drawn, and analyzed for A1c levels and albumin levels. During the first, fourth, eighth, and sixteenth week, following Saliva-Check BUFFER Kit testing done before HBO therapy, additional saliva will be collected to ensure that a minimum of 2 mL of saliva can be stored at less than or equal to -20 oC for protein analysis.

After salivary testing, each patient will enter a hyperbaric oxygen chamber located at Loma Linda University Medical Center. The patient will gradually be elevated to therapeutic oxygen levels over an 8-12 minute period. At this time, 100% oxygen will be administered at 2.0 ATA or 2.5 ATA, at the discretion of the treating physician, for 90 minutes. A 10-minute air-break will be given after the first 45 minutes if the patients are on the 2.5 ATA protocol. At the conclusion of the oxygen treatment, the oxygen and pressure levels are gradually decreased over 8-12 minutes to return to a depth of 1 ATA. After exiting the hyperbaric oxygen chamber, salivary testing will once again be performed on each patient.

Collected data will be compared to two independent control groups. The Positive Control Group will include 26 individuals who fit the inclusion and exclusion criteria: participants for whom hyperbaric oxygen treatment is indicated, but who have not had radiation therapy for head or neck cancer. The Negative Control Group will include the first 26 individuals who fit the inclusion and exclusion criteria: participants who have previously had head and neck radiation therapy, but for whom hyperbaric oxygen treatment is not indicated. Salivary data for the Positive Control Group will be collected in such as way as to parallel data collected for the Treatment Group. Salivary data will be collected in the same way for the Negative Control Group with the following modifications: salivary flow rate testing will only be performed once during each visit and salivary testing will be spaced on the basis of time in days in contrast to number of hyperbaric oxygen treatment sessions.

ELIGIBILITY:
Inclusion Criteria:

* Patient age: 18+.
* Patient must give informed consent.

Treatment Group

* Patient has completed head and neck irradiation treatment.
* Hyperbaric oxygen therapy is indicated and patient has accepted said treatment.
* Patient must be able to complete hyperbaric oxygen course of treatment.

Positive Control Group

* Hyperbaric oxygen therapy is indicated and patient has accepted said treatment.
* Patient must be able to complete hyperbaric oxygen course of treatment.

Negative Control Group

* Patient has completed head and neck irradiation treatment.
* Hyperbaric oxygen therapy has not been used.

Exclusion Criteria:

* Currently using anti-cholinergic agent, eg: Scopolamine patch, Atropine, Ipratropium, Spiriva.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the Loma Linda University Healthcare System
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-08; Primary Completion 2021-08 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Volume of Stimulated Saliva | Pre-treatment to post treatment, average duration of 12 weeks

SECONDARY OUTCOMES:
Concentrations of Salivary Thrombospondin-1 | Measured weekly, average duration of treatment is 12 weeks
  Measurements will occur at baseline and weekly throughout treatment with one post treatment measurement one week after last treatment
Concentration of Salivary IGF-1 | Measured weekly, average duration of treatment is 12 weeks
  Measurements will occur at baseline and weekly throughout treatment with one post treatment measurement one week after last treatment
Concentration of Salivary VEGF-A | Measured weekly, average duration of treatment is 12 weeks
  Measurements will occur at baseline and weekly throughout treatment with one post treatment measurement one week after last treatment
Salivary pH | Measured weekly, average duration of treatment is 12 weeks
  Measurements will occur at baseline and weekly throughout treatment with one post treatment measurement one week after last treatment
Salivary buffering capacity | Measured weekly, average duration of treatment is 12 weeks
  Measurements will occur at baseline and weekly throughout treatment with one post treatment measurement one week after last treatment
Impact of HBO treatment on quality of life for ORN patients with xerostomia | Pre to Post Treatment, average duration of treatment is 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Takkin Lo, MD, MPH, Principal Investigator — Loma Linda University School of Medicine
Locations (1):
- Loma Linda University Health System, Loma Linda, California, United States